CLINICAL TRIAL: NCT05334563
Title: The Incidence of Congenital Combined Pituitary Hormone Deficiency in Denmark - a National Observational Study
Brief Title: Incidence of cCPHD in Denmark - a National Observational Study
Acronym: IcCPHD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Christesen, Clinical professor of Medicine, Odense University Hospital
Other Study IDs: IcCPHD
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Combined Pituitary Hormone Deficiency Genetic Form; Combined Pituitary Hormone Deficiency
Keywords: Combined pituitary hormone deficiency; Congenital combined pituitary hormone deficiency; Congenital multiple pituitary hormone deficiency; Incidence of pituitary hormone deficiency
MeSH Terms: conditions — Combined Pituitary Hormone Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The pituitary gland is a small pea-sized gland that produces a variety of important hormones. Some children are born with a deficient production of two or more pituitary hormones. This rare and potentially severe disease is called congenital combined pituitary hormone deficiency (cCPHD).

cCPHD can cause many different symptoms, some of which appear shortly after birth and others later in childhood. Symptoms that appear shortly after birth are e.g., development of very low blood sugar, disturbances in the salt balance, and severe dehydration, whereas symptoms that appear later in life are short stature, missing pubertal development, fatigue, and sensitiveness to cold. Fortunately, it is possible to replace the missing hormones.

Currently, it is unknown how common cCPHD is. Therefore, the investigators wish to examine 1) how many children are diagnosed with cCPHD before the age of 18 years, 2) how many children are diagnosed with cCPHD at age <1 year, 1-8 years, 9-17 years, and 3) the patients' hormone deficiency characteristics and brain MRI scans.

The investigators will identify the patients by searching for diagnosis codes used for pituitary disease and pituitary malformations in the Danish National Patient Registry and locally at the four hospitals approved for the treatment of cCPHD in children. Through the searches, the investigators expect to identify approximately 1500 patients. The investigators will then review the hospital files of all identified patients to exclude patients with only one hormone deficiency and patients with an acquired cause of the disease. The investigators aim to include all cCPHD patients in Denmark born in the period 1996 and 2020.

DETAILED DESCRIPTION:
1. Background

   Congenital combined pituitary hormone deficiency (cCPHD) is defined as the partial or complete loss of more than one hormone secreted from the pituitary gland, caused by genetic or prenatal factors. Combined pituitary hormone deficiency (CPHD) is a broader term covering both congenital and acquired forms.

   The incidence and prevalence of cCPHD are not known.

   Pituitary hormone deficiencies most commonly occur in the adenohypophysis involving growth hormone (GH), thyroid-stimulating hormone (TSH), corticotropin (ACTH), prolactin, luteinizing hormone (LH) and follicle-stimulating hormone (FSH). More rarely, the neurohypophysis is also affected, resulting in vasopressin deficiency.

   Symptoms and clinical features of cCPHD are variable, even within the same family, including the extent and severity of the hormone deficiencies, the age of clinical onset and the cerebral comorbidity. Moreover, delay inadequate treatment may affect the clinical outcome and prognosis.

   Newborns with clinical overt cCPHD may present in the first days of life with hypoglycemia, electrolyte abnormalities, hypothermia, conjugated hyperbilirubinemia, poor appetite, vomiting, and failure to thrive. In boys, gonadotropin deficiency may present with hypogonadism including micropenis. Patients with vasopressin deficiency may have central diabetes insipidus from birth with polyuria and quickly develop severe hypernatremic dehydration.

   Delayed onset of cCHPD may occur as a gradual process, usually with growth hormone deficiency (GHD) as the first manifestation, followed by TSH deficiency and later other hormone deficiencies including FSH/LH deficiency.

   MRI of the brain and the pituitary region commonly, but not always, reveal anatomical abnormalities including aplasia or hypoplasia of the adenohypophysis and/or pituitary stalk. Aplasia, hypoplasia, or ectopic position of the neurohypophysis may be seen. Associated brain abnormalities may include septo-optic dysplasia (SOD) and aplasia/hypoplasia of other brain structures, especially in the midline. Syndromes, including cCPHD with other brain or organ abnormalities, include heterotaxy syndrome, Worster-Drought Syndrome, congenital proprotein convertase 1/3 deficiency, FOXA2 mutation syndrome and many others.

   Genetic testing can be helpful to understand the diverse phenotypic picture of cCPHD.

   The development of the pituitary gland is dependent on the sequential temporal and spatial expression of transcription factors and signaling molecules and occurs in a well-defined sequence of events. Some of these factors include HESX1, LHX3, LHX4, POU1F1, PROP1, SIX6, OTX2, PITX2, GLI2, and SOX3, all of which have been shown to play a role in the development and maturation of the pituitary gland.

   Disruption of this cascade due to mutations in any of these gene products affects the ontogeny of one or several of the pituitary cell types and ultimately leads to hormone deficiency with or without extra-pituitary abnormalities. Previous studies have shown a higher prevalence of genetic mutations in familial cases, where both dominant, recessive and X-linked inheritance has been demonstrated. Still, most patients with cCPHD have remained genetically unexplained.

   The treatment of cCPHD consists of the substitution of the deficient pituitary hormones or their target hormones, including growth hormone, thyroid hormone, sex hormones, glucocorticoids, and vasopressin. Eventual other cerebral or other organ syndromal manifestations must be identified and managed.
2. Materials and methods

   This study is a national study based on ICD10 diagnosis codes from The Danish National Patient Registry (DNPR) and the four tertiary hospitals: Odense Universitetshospital, Aarhus Universitetshospital, Rigshospitalet, and Aalborg Universitetshospital. The DNPR contains a unique registration of all hospitalized patients in the country since 1977; with WHO ICD10 diagnosis codes since 1994. The registry identifies patients based on the unique personal identification number of each person living in Denmark. The diagnosis code searches at the four tertiary hospitals are made in addition to the DNPR search to provide a higher probability of identifying all patients with cCPHD in Denmark.

   The DNPR and the four local hospital searches will be performed using the ICD10 codes E23.0-E23.9 (pituitary hormone deficiencies and other diseases in the pituitary gland), Q89.2G (congenital malformation of the pituitary), and Q04.0-Q04.9 (other congenital brain malformations) for the 25-year period: 1st of January 1996 - 31st of December 2020. Patients with the additional diagnoses C69.0-C72.9 (cancer in eyes, brain, other parts of the CNS), C75.1-C75.3 (cancer in the pituitary, corpus pinealis and craniopharyngeomas), D35.2 - D35.4 (benign tumours of the pituitary gland, corpus pineale, or ductus craniopharyngei) and D33.0-D33.9 (benign tumours in the brain and spinal cord) will be excluded. Patients with the ICD10 diagnosis codes A80.0-A89.9 (central nervous system infections) and/ or I60.0-I64.9 (nontraumatic subarachnoid hemorrhage, nontraumatic intracerebral hemorrhage, other and unspecified nontraumatic intracranial hemorrhage, cerebral infarction, stroke not specified as haemorrhage or infarction) registered before the time of the E23.0-E23.9 diagnosis will also be excluded.

   For the identified patients a retrospective hospital file review will be performed to confirm the cCPHD diagnosis and to exclude patients who meet one of the exclusion criteria.

   The data used in this project are found in patient journals and include the following: birthdate, sex as indicated by the presence of male/female genitals (male/female), born in Denmark (yes/no), presence of ICD-10 diagnosis codes of interest (yes/no), date and results of blood samples and stimulation tests of interest (low/normal/inadequately high/high), date and result of urine osmolality measurement (low/normal/high), abnormalities of the adenohypophysis, neurohypophysis, pituitary stalk, midline and cerebrum by the latest MRI (aplasia/hypoplasia/ectopic/normal or yes/no), and hospital file descriptions of clinical features of hormone deficiencies (yes/no).

   All hormone deficiencies will be retrospectively validated using a set of hormone deficiency criteria. The criteria were defined by five experienced pediatric endocrinologists, including a representative from each of the highly specialized hospitals, and were based on national and international endocrinological guidelines, published literature, and the clinical practice at the highly specialized hospitals.
3. Ethics

   This study was approved by the Management Secretariat and the Regional Secretariat and Law of The Region of Southern Denmark (j.no. 20/58158). To ensure compliance with The General Data Protection Regulation and The Danish Data Protection Act, data were collected and managed in collaboration with Open Patient data Explorative Network (OPEN) using Microsoft SharePoint and REDCap (Research Electronic Data Capture).
4. Participatory design

   The study protocol is designed after preliminary contacts with 10 parents to children with cCPHD at Odense University Hospital. The parents expressed a need of dissemination of several aspects of cCPHD to improve future management of this rare disease. Some stressed the need of identification of early signs of cCPHD to contribute to fastest possible diagnosis, as diagnosis delay has been a major, sometimes life-threatening problem for their children, e.g. severe hypernatriemic dehydration with a s-sodium of 180 mmol/L in a neonate with cCPHD and diabetes insipidus. Others stressed the benefits of dissemination of good results of early and centralized expert treatment including androgen therapy in infant boys with hypogonadism. Others wanted to pass on a message that children with non-syndromic cCPHD can live a normal life with normal school performance. Others stressed that CPHD should be looked for in syndromes with potential CPHD or children with an unknown syndrome to optimize e.g. their growth and cerebral function. One parent has agreed to be a part of the project group.
5. Perspectives

   Given that cCPHD is a rare and complex, potentially life-threatening disease, the paucity of literature on the subject and the lack of estimates of incidence, this study is expected to provide important information to be published. A good understanding of the illness is crucial and may lead to patients getting diagnosed earlier.
6. Dissemination of the results

   The study will be published as one or two papers in peer-reviewed international journals. A Danish and English press release will be made at the time of publication. Oral presentation(s) or poster(s) will be presented at national meetings, e.g. The Danish Society of Paediatric Endocrinology (DSPE) and international meetings, e.g. the annual European Society of Paediatrics (ESPE) meeting or ENDO. A popular talk is scheduled at a meeting in patient organization The Danish Pituitary Network
7. Project group

   Henrik Thybo Christesen, Consultant, Professor, ph.d, MD, Hans Christian Andersen Children's Hospital, Odense University Hospital, Denmark. Project supervisor.

   Dorte Hansen, Consultant, Associate Professor, ph.d, MD, Hans Christian Andersen Children's Hospital, Odense University Hospital, Denmark. Project co-supervisor.

   Niels Holtum Birkebæk, Consultant, ph.d, MD, Dept. of Pediatrics, Aarhus University Hospital Skejby, Denmark. Study site collaborator.

   Ann-Margrethe Rønholt Christensen, Associate professor, Dept. of Pediatrics, Aalborg University Hospital, Denmark. Study site collaborator.

   Rikke Bodin Beck-Jensen, Consultant, ph.d, MD, Dept. Of Growth and Reproduction, Rigshospitalet. Study site collaborator

   Louise Kjersgaard Jakobsen, research year medical student
8. Fonds

This work was supported by Odense University Hospital Fund (j.no. A4599), and Dagmar Marshalls Fund (29/04/2021).

ELIGIBILITY:
Inclusion Criteria:

* Born between January 1, 1996, and December 31, 2020.
* Registered in Danish National Patient Registry or locally at Hans Christian Andersen Children´s Hospital, Odense University Hospital, Department of Growth and Reproduction, Rigshospitalet, Department of Pediatrics and Adolescent Medicine, Aarhus University Hospital or Department of Pediatrics, Aalborg University Hospital with an ICD-10 diagnosis code E23·0-E23·9 (hypofunction and other disorders of pituitary) and/or Q89·2G (congenital malformation of pituitary) before age 15 years.
* Validated secondary/tertiary deficiency of two pituitary hormones before age 18 years.

Exclusion Criteria:

* ICD-10 diagnosis codes indicating acquired PHD.
* No available hospital files.
* Less than two documented secondary/tertiary hormone deficiencies.
* Acquired CPHD.

Ages: 1 Day to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study aims to include all congenital combined pituitary hormone deficiency patients in Denmark born between January 1, 1996, and December 31, 2020, identified through the ICD-10 diagnosis code searches in the Danish National Patient Registry and locally at the four highly specialized hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of congenital combined pituitary hormone deficiency in Denmark diagnosed before age 18 years. | 1996 to 2020
  Incidence per 100.000 live births and incidence rate per 1 million live births per year

SECONDARY OUTCOMES:
The incidence of congenital combined pituitary hormone deficiency in Denmark diagnosed at age <1 year, 1-8 years, and 9-17 years. | 1996 to 2020
  Incidence per 100.000 live births and incidence rate per 1 million live births per year
Hormone deficiency characteristics and brain MRI abnormalities in the congenital combined pituitary hormone deficiency patients | 1996 to 2020
  Abnormalities of the adenohypophysis, neurohypophysis, pituitary stalk, midline and cerebrum by the latest MRI (aplasia/hypoplasia/ectopic/normal or yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik T Christesen, ph.d., Principal Investigator — Hans Christian Andersen Children´s Hospital, Odense University Hospital
Locations (1):
- HCA Research, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The de-identified patient data that underlie this study are available to researchers upon approval by the Region of Southern Denmark. The study protocol and the Stata do-files are available to anyone with a request.
Supporting Information: Study Protocol
Time Frame: Proposals can be submitted up to three years following article publication and should be directed to henrik.christesen@rsyd.dk.
Access Criteria: Approval by the Region of Southern Denmark.

REFERENCES:
- [Background] Romero CJ, Nesi-Franca S, Radovick S. The molecular basis of hypopituitarism. Trends Endocrinol Metab. 2009 Dec;20(10):506-16. doi: 10.1016/j.tem.2009.06.005. Epub 2009 Oct 23. PMID 19854060
- [Background] Romero CJ, Pine-Twaddell E, Radovick S. Novel mutations associated with combined pituitary hormone deficiency. J Mol Endocrinol. 2011 Jun 9;46(3):R93-R102. doi: 10.1530/JME-10-0133. Print 2011 Jun. PMID 21447626
- [Background] Choi JH, Jung CW, Kang E, Kim YM, Heo SH, Lee BH, Kim GH, Yoo HW. Rare Frequency of Mutations in Pituitary Transcription Factor Genes in Combined Pituitary Hormone or Isolated Growth Hormone Deficiencies in Korea. Yonsei Med J. 2017 May;58(3):527-532. doi: 10.3349/ymj.2017.58.3.527. PMID 28332357
- [Background] Haim-Pinhas H, Kauli R, Lilos P, Laron Z. Growth, development, puberty and adult height of patients with congenital multiple pituitary hormone deficiencies. Growth Horm IGF Res. 2016 Apr;27:46-52. doi: 10.1016/j.ghir.2016.01.004. Epub 2016 Feb 19. PMID 26947989
- [Background] Di Iorgi N, Morana G, Allegri AE, Napoli F, Gastaldi R, Calcagno A, Patti G, Loche S, Maghnie M. Classical and non-classical causes of GH deficiency in the paediatric age. Best Pract Res Clin Endocrinol Metab. 2016 Dec;30(6):705-736. doi: 10.1016/j.beem.2016.11.008. Epub 2016 Nov 24. PMID 27974186
- [Background] de Graaff LC, Argente J, Veenma DC, Drent ML, Uitterlinden AG, Hokken-Koelega AC. PROP1, HESX1, POU1F1, LHX3 and LHX4 mutation and deletion screening and GH1 P89L and IVS3+1/+2 mutation screening in a Dutch nationwide cohort of patients with combined pituitary hormone deficiency. Horm Res Paediatr. 2010;73(5):363-71. doi: 10.1159/000308169. Epub 2010 Apr 14. PMID 20389107
- [Background] De Rienzo F, Mellone S, Bellone S, Babu D, Fusco I, Prodam F, Petri A, Muniswamy R, De Luca F, Salerno M, Momigliano-Richardi P, Bona G, Giordano M; Italian Study Group on Genetics of CPHD. Frequency of genetic defects in combined pituitary hormone deficiency: a systematic review and analysis of a multicentre Italian cohort. Clin Endocrinol (Oxf). 2015 Dec;83(6):849-60. doi: 10.1111/cen.12849. Epub 2015 Aug 6. PMID 26147833
- [Background] Kelberman D, Rizzoti K, Lovell-Badge R, Robinson IC, Dattani MT. Genetic regulation of pituitary gland development in human and mouse. Endocr Rev. 2009 Dec;30(7):790-829. doi: 10.1210/er.2009-0008. Epub 2009 Oct 16. PMID 19837867
- [Background] Brodsky MC, Conte FA, Taylor D, Hoyt CS, Mrak RE. Sudden death in septo-optic dysplasia. Report of 5 cases. Arch Ophthalmol. 1997 Jan;115(1):66-70. doi: 10.1001/archopht.1997.01100150068011. PMID 9006427
- [Background] Cameron FJ, Khadilkar VV, Stanhope R. Pituitary dysfunction, morbidity and mortality with congenital midline malformation of the cerebrum. Eur J Pediatr. 1999 Feb;158(2):97-102. doi: 10.1007/s004310051026. PMID 10048603
- [Background] Child CJ, Blum WF, Deal C, Zimmermann AG, Quigley CA, Drop SL, Cutler GB Jr, Rosenfeld RG. Development of additional pituitary hormone deficiencies in pediatric patients originally diagnosed with isolated growth hormone deficiency due to organic causes. Eur J Endocrinol. 2016 May;174(5):669-79. doi: 10.1530/EJE-15-1203. Epub 2016 Feb 17. PMID 26888628
- [Background] Cerbone M, Dattani MT. Progression from isolated growth hormone deficiency to combined pituitary hormone deficiency. Growth Horm IGF Res. 2017 Dec;37:19-25. doi: 10.1016/j.ghir.2017.10.005. Epub 2017 Oct 19. PMID 29107171
- [Background] Ascoli P, Cavagnini F. Hypopituitarism. Pituitary. 2006;9(4):335-42. doi: 10.1007/s11102-006-0416-5. PMID 17077946
- [Background] Braslavsky D, Keselman A, Chiesa A, Bergada I. [Diagnosis of congenital endocrinological disease in newborns with prolonged jaundice and hypoglycaemia]. An Pediatr (Barc). 2012 Mar;76(3):120-6. doi: 10.1016/j.anpedi.2011.08.011. Epub 2011 Oct 20. Spanish. PMID 22015010
- [Background] Toogood AA, Stewart PM. Hypopituitarism: clinical features, diagnosis, and management. Endocrinol Metab Clin North Am. 2008 Mar;37(1):235-61, x. doi: 10.1016/j.ecl.2007.10.004. PMID 18226739
- [Derived] Jakobsen LK, Jensen RB, Birkebaek NH, Hansen D, Christensen AR, Bjerrum MC, Christesen HT. Diagnosis and Incidence of Congenital Combined Pituitary Hormone Deficiency in Denmark-A National Observational Study. J Clin Endocrinol Metab. 2023 Sep 18;108(10):2475-2485. doi: 10.1210/clinem/dgad198. PMID 37043518

DOCUMENTS (1):
  • Study Protocol (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT05334563/Prot_001.pdf